CLINICAL TRIAL: NCT03311425
Title: The Effects of Intraoperative Local and Systemic Corticosteroid Administration on Postoperative Dysphagia After Anterior Cervical Fusion
Brief Title: Effect of Local Intraoperative Steroid on Dysphagia After ACDF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Kern Singh, Professor of Orthopaedic Surgery, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13092002
Record Dates: First submitted 2017-10-09; First posted 2017-10-17 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Dysphagia
Keywords: Anterior cervical discectomy and fusion; prevertebral swelling; swallowing; methylprednisolone; intraoperative steroid
MeSH Terms: conditions — Deglutition Disorders | interventions — Methylprednisolone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Depomedrol plus IV dexamethasone (Active Comparator): Local intraoperative application of methylprednisolone (Depomedrol) plus standard systemic (IV) dexamethasone
  Interventions: Drug: Methylprednisolone; Drug: Dexamethasone
- IV dexamethasone (Placebo Comparator): Intraoperative systemic (IV) steroid (dexamethasone) only.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Methylprednisolone — Application of 40mg Depomedrol (methylprednisolone acetate) suspension into the retropharyngeal space prior to incision closure
  Arms: Local Depomedrol plus IV dexamethasone
Drug: Dexamethasone — Administration of 10mg Dexamethasone IV intraoperatively

SUMMARY:
The purpose of this study is to determine if the incidence and duration of postoperative dysphagia are improved in the participants receiving a local injection of methylprednisolone with systemic dexamethasone when compared to those receiving the usual systemic dexamethasone.

DETAILED DESCRIPTION:
Postoperative dysphagia is a known complication of anterior cervical spinal fusion (ACF) surgery with a published incidence that ranges from 1.7% to 50.3%.1-9 The pathophysiology of post-operative dysphagia is not fully understood and is subject to further study. Postoperative dysphagia has been reported to improve with time with a mean incidence of 19.8% at 6 months, 16.8% at 12 months, and 12.9% at 24 months after ACDF. The investigator's standard of practice is to provide 10mg of dexamethasone IV intraoperatively in order to reduce postoperative prevertebral soft tissue swelling. Despite the growing popularity of ACDF procedures, there is a lack of clear evidence supporting the utilization of perioperative corticosteroids in the setting of an ACDF.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary 1- to 3-level ACDF:

  (a) Diagnosis: myelopathy, radiculopathy, myeloradiculopathy, stenosis, herniated nucleus pulposus, degenerative disc disease, spondylosis, osteophytic complexes, and foraminal stenosis
* Patients able to provide informed consent

Exclusion Criteria:

* Allergies or other contraindications to medicines in the protocol including:

  (a) Existing history gastrointestinal bleeding
* Existing history of dysphagia
* Current Smokers
* Cervical spine trauma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline SWAL-QOL survey at 3 months | 3 months
  In the postoperative period, patients will be asked to complete the SWAL-QOL survey at the 3 month follow up office visit. This will be compared to preoperative scores. Each survey is scored out of 100 with minimum score of 20 indicating severe dysphagia and 100 indicating no dysphagia/normal swallowing. As such, a greater decrease in SWAL-QOL score from preoperative (baseline) to 3 month visit indicates greater postoperative swallowing difficulty.

SECONDARY OUTCOMES:
Change from Baseline Prevertebral Soft Tissue Swelling at 3 months | 3 months
  Prevertebral soft tissue swelling will be measured utilizing the standard of practice plain lateral radiographs that are obtained at the 3 month postoperative follow up office visit.The area of the prevertebral soft tissue density will be measured from the caudal border of C1 to the cranial end plate of C7 with a digital measuring instrument. These measurements will be compared to the preoperative measurements obtained utilizing the preoperative lateral plain radiographs which are also standard of practice.
Adverse Events | 1 year
  Any perioperative or postoperative adverse events will be recorded and evaluated between cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Kern Singh, MD, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caspar W, Barbier DD, Klara PM. Anterior cervical fusion and Caspar plate stabilization for cervical trauma. Neurosurgery. 1989 Oct;25(4):491-502. doi: 10.1097/00006123-198910000-00001. PMID 2797387
- [Background] Saunders RL, Bernini PM, Shirreffs TG Jr, Reeves AG. Central corpectomy for cervical spondylotic myelopathy: a consecutive series with long-term follow-up evaluation. J Neurosurg. 1991 Feb;74(2):163-70. doi: 10.3171/jns.1991.74.2.0163. PMID 1988583
- [Background] Stewart M, Johnston RA, Stewart I, Wilson JA. Swallowing performance following anterior cervical spine surgery. Br J Neurosurg. 1995;9(5):605-9. doi: 10.1080/02688699550040882. PMID 8561932
- [Background] Martin RE, Neary MA, Diamant NE. Dysphagia following anterior cervical spine surgery. Dysphagia. 1997 Winter;12(1):2-8; discussion 9-10. doi: 10.1007/pl00009513. PMID 8997826
- [Background] Schneeberger AG, Boos N, Schwarzenbach O, Aebi M. Anterior cervical interbody fusion with plate fixation for chronic spondylotic radiculopathy: a 2- to 8-year follow-up. J Spinal Disord. 1999 Jun;12(3):215-20; discussion 221. PMID 10382774
- [Background] Frempong-Boadu A, Houten JK, Osborn B, Opulencia J, Kells L, Guida DD, Le Roux PD. Swallowing and speech dysfunction in patients undergoing anterior cervical discectomy and fusion: a prospective, objective preoperative and postoperative assessment. J Spinal Disord Tech. 2002 Oct;15(5):362-8. doi: 10.1097/00024720-200210000-00004. PMID 12394659
- [Background] Bazaz R, Lee MJ, Yoo JU. Incidence of dysphagia after anterior cervical spine surgery: a prospective study. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2453-8. doi: 10.1097/00007632-200211150-00007. PMID 12435974
- [Background] Smith-Hammond CA, New KC, Pietrobon R, Curtis DJ, Scharver CH, Turner DA. Prospective analysis of incidence and risk factors of dysphagia in spine surgery patients: comparison of anterior cervical, posterior cervical, and lumbar procedures. Spine (Phila Pa 1976). 2004 Jul 1;29(13):1441-6. doi: 10.1097/01.brs.0000129100.59913.ea. PMID 15223936
- [Background] Yue WM, Brodner W, Highland TR. Persistent swallowing and voice problems after anterior cervical discectomy and fusion with allograft and plating: a 5- to 11-year follow-up study. Eur Spine J. 2005 Sep;14(7):677-82. doi: 10.1007/s00586-004-0849-3. Epub 2005 Feb 4. PMID 15692825
- [Background] Lee JY BR, Furey CG, ., et al. Dysphagia after anterior cervical spine surgery: Pathophysiology, incidence, and prevention. Cervical Spine Research Society 2007.
- [Background] Lee MJ, Bazaz R, Furey CG, Yoo J. Risk factors for dysphagia after anterior cervical spine surgery: a two-year prospective cohort study. Spine J. 2007 Mar-Apr;7(2):141-7. doi: 10.1016/j.spinee.2006.02.024. Epub 2007 Jan 22. PMID 17321961
- [Background] Riley LH 3rd, Skolasky RL, Albert TJ, Vaccaro AR, Heller JG. Dysphagia after anterior cervical decompression and fusion: prevalence and risk factors from a longitudinal cohort study. Spine (Phila Pa 1976). 2005 Nov 15;30(22):2564-9. doi: 10.1097/01.brs.0000186317.86379.02. PMID 16284596
- [Background] Lee MJ, Bazaz R, Furey CG, Yoo J. Influence of anterior cervical plate design on Dysphagia: a 2-year prospective longitudinal follow-up study. J Spinal Disord Tech. 2005 Oct;18(5):406-9. doi: 10.1097/01.bsd.0000177211.44960.71. PMID 16189451
- [Background] Vaidya R, Carp J, Sethi A, Bartol S, Craig J, Les CM. Complications of anterior cervical discectomy and fusion using recombinant human bone morphogenetic protein-2. Eur Spine J. 2007 Aug;16(8):1257-65. doi: 10.1007/s00586-007-0351-9. Epub 2007 Mar 27. PMID 17387522
- [Background] Riley LH 3rd, Vaccaro AR, Dettori JR, Hashimoto R. Postoperative dysphagia in anterior cervical spine surgery. Spine (Phila Pa 1976). 2010 Apr 20;35(9 Suppl):S76-85. doi: 10.1097/BRS.0b013e3181d81a96. PMID 20407354
- [Background] Pedram M, Castagnera L, Carat X, Macouillard G, Vital JM. Pharyngolaryngeal lesions in patients undergoing cervical spine surgery through the anterior approach: contribution of methylprednisolone. Eur Spine J. 2003 Feb;12(1):84-90. doi: 10.1007/s00586-002-0495-6. Epub 2002 Dec 4. PMID 12592551
- [Background] Nam TW, Lee DH, Shin JK, Goh TS, Lee JS. Effect of intravenous dexamethasone on prevertebral soft tissue swelling after anterior cervical discectomy and fusion. Acta Orthop Belg. 2013 Apr;79(2):211-5. PMID 23821974
- [Derived] Haws BE, Khechen B, Narain AS, Hijji FY, Bohl DD, Massel DH, Mayo BC, Ahn J, Singh K. Impact of local steroid application on dysphagia following an anterior cervical discectomy and fusion: results of a prospective, randomized single-blind trial. J Neurosurg Spine. 2018 Jul;29(1):10-17. doi: 10.3171/2017.11.SPINE17819. Epub 2018 Apr 20. PMID 29676673